CLINICAL TRIAL: NCT02113215
Title: Very Low Density Lipoprotein Turnover in Young and Elderly Individuals
Status: Terminated | Type: Observational
Why Stopped: PI left UTMB
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 11-318; 1R01AG033761-01A1 (NIH)
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Aging
Keywords: aging; lipid metabolism; very low density lipoproteins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and muscle biopsies will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Young Males: Males, age 18-35 years. 9-hour Stable isotope infusion
  Interventions: Procedure: Stable Isotope Infusion
- Young Females: Females, age 18-35 years. 9-hour Stable isotope infusion
  Interventions: Procedure: Stable Isotope Infusion
- Older Males: Males, age 60-75. 9-hour Stable isotope infusion
  Interventions: Procedure: Stable Isotope Infusion
- Older Females: Females, age 60-75. 9-hour Stable isotope infusion
  Interventions: Procedure: Stable Isotope Infusion

INTERVENTIONS:
Procedure: Stable Isotope Infusion — 9-hour infusion of stable isotope tracers

SUMMARY:
Intrahepatic and intramyocellular lipid concentrations are elevated in elderly individuals relative to young people, despite no significant difference in fasting plasma TAG concentrations. Our general hypothesis is that the increase in intrahepatic fat with age results from reduced VLDL turnover, and therefore elderly individuals in this study will display lower VLDL turnover rates than young individuals. The aims of this study are a) to compare VLDL turnover in young and elderly individuals, and b) to compare a bolus method and a constant infusion method of assessing VLDL turnover.

DETAILED DESCRIPTION:
Several studies have shown an association between hypertriacylglycerolaemia and coronary artery disease. Additionally, ectopic fat distribution, in particular, deposition of excess lipid within the liver and skeletal muscle, has been shown to correlate negatively with insulin sensitivity, thus presenting a metabolic milieu in which risk of developing type 2 diabetes is elevated. Previous research from our group has shown that the triacylglycerol (TAG) concentration within the liver, and within skeletal muscle fibres IMCLs (intramyocellular lipids), is increased in elderly individuals compared with young people. The elevation of lipids in these particular tissues for the elderly group was observed despite no statistically significant difference in fasting plasma TAG concentration. As the plasma TAG concentration during the postabsorptive state is largely determined by the production and clearance rates of very low density lipoprotein triacylglycerol (VLDL-TAG), and increased liver fat content has been shown to drive production of large VLDL particles, it is important to gain an understanding of whether VLDL synthesis and breakdown differs between young and elderly individuals. Such new knowledge may offer an insight into why tissue lipids are elevated in the elderly. At present, no data exist in the literature describing VLDL turnover in elderly people. We hypothesise that very low density lipoprotein turnover will be reduced in elderly individuals compared with young people. The aims of this study are a) to determine whether fractional synthesis and breakdown rates of both the protein and lipid parts of the VLDL are different between young and elderly individuals, and b) to determine whether VLDL turnover values appear different when calculated using a constant infusion tracer method as compared with a bolus tracer method. Eight young men, eight young women, eight elderly men and eight elderly women will each participate in an 8-hour infusion study. Stable isotopes of glycerol, amino acids and fatty acids will be infused, and blood samples will be drawn in intervals during the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 35 years, or 60 to 75 years.
* Body mass index ≤ 27 kg•m2
* Ability to sign informed consent.
* Score of ≥26 for Mini-Mental State Exam

Exclusion Criteria:

* Diabetics (plasma glucose concentration >200 mg/dl at 2 hr after oral intake of 75 g glucose).
* Fasting plasma triacylglycerol concentration above 500 mg/dl
* Kidney disease.
* Liver disease.
* Bleeding disorders.
* Anaemia (Hb < 13 g/dl in males or < 12 g/dl in females).
* Endocrine disease (with the exception of well-regulated hypothyroidism).
* Positive hepatitis or HIV screens.
* Alcohol (CAGE questionnaire; abnormal liver enzyme values) or drug abuse (amphetamines, cocaine, opioids, marijuana).
* Lipid altering agents.
* Score of <26 for Mini-Mental State Exam

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals from the Galveston area.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Very Low Density Lipoprotein (VLDL) Turnover | 9-hours
  Turnover rates of VLDL-triglycerides and VLDL-ApoB (apolipoprotein B)-100, including synthesis and breakdown rates, measured during a 9-hour infusion trial.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Borsheim, Ph.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Dept of Surgery, Galveston, Texas, United States